CLINICAL TRIAL: NCT03958266
Title: A Feasibility Study of a Novel Mobile Phone Application in the Long Term Management of Patients With Inflammatory Bowel Diseases
Brief Title: MyIBD Care - Feasibility Study
Status: Withdrawn | Type: Observational
Why Stopped: COVID pandemic
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 266567
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2019-05

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MyIBD Care - Study Group: Will have traditional face to face outpatient contacts replaced with a novel mobile phone application supported via a digital clinician portal
  Interventions: Device: MyIBD Care

INTERVENTIONS:
Device: MyIBD Care — Novel mobile phone application

SUMMARY:
The aim of this study is appraise the safety and feasibility of utilising a novel mobile phone application and linked clinical platform to replace and enhance traditional outpatient appointments for patients with Inflammatory Bowel Diseases. The goal of this study is to demonstrate whether the platform can reduce the costs of managing patients on complex immunomodulators and biologic therapies whilst maintaining safety monitoring such as clinical patient reported outcome measures (PROMs), haematological and biochemical tests.

DETAILED DESCRIPTION:
15 million people in the England suffer from long term conditions (LTCs). Furthermore, the number of people with three or more LTC's has risen from 1.9 million people in 2008 to 2.9 million in 2018. And with the growing number of people suffering from these conditions, the pressure grows for health care providers to provide long term solutions to meet this increase in demand.

Inflammatory Bowel Disease (IBD) is an exemplar for LTCs, requiring frequent routine appointments, an ongoing testing regimen and costly pharmacological intervention. Moreover, people living with Crohn's disease (CD) or Ulcerative Colitis (UC) are often young and report that their condition leads to a significant reduction in quality of life (QOL) even when symptoms are relatively well-controlled. Patients present with diarrhoea, abdominal pain, weight loss and other symptoms that have a significant impact on quality of life (taking into account social functioning, employment status, psychological distress). The condition has an estimated prevalence of 0.3% in North America, Northern Europe and Oceania (1) with a substantial direct and indirect costs. The majority of patients require lifelong medication and are followed up in secondary care. Like many immune mediated inflammatory conditions, it is a disease of relapse and remission. At times of relapse patients require rapid access to specialist advice, managing flares early leads to better outcomes such as returning to work or daily activities and avoids costly admission to hospital.

Up to 76% of patients with CD and 51% with UC, will need immunomodulators (thiopurines or methotrexate) which require regular blood monitoring at minimum 4 times per year to screen for side effects of myeloid and hepatotoxicity (2). Patients on sub-cutaneous biologic medications such as adalimumab, golimumab and Ustekinumab also require regular blood monitoring which often necessitates clinic visits. In a recent nationwide survey of 2400 consecutive outpatient appointments in a wide variety of hospitals throughout England and Scotland up to 75% of patients were deemed to be in a quiescent or mildly active phase of disease (2). The majority of those patients are being seen in outpatients based on an antiquated model of routine follow up appointments, with dates of 2, 3, 4, 6 and 12-month intervals chosen either to have safety-based blood tests or a date arbitrarily chosen by clinician or patient. Appointments such as these rarely reflect a clinical need and lead to an inflexible system in which patients Clinicians at King's College Hospital wanted to explore whether digital self-management could be an effective way of reducing the burden the condition places on the patient and on the health system. Using the My IBD Care app, they provided patients with a convenient digital touchpoint for their treatment, facilitating easy access to information, including their care plan, health record and self-management content; and digital contact with hospital staff via an app.

From a hospital perspective, self-managing patients cost less to treat and place less of a burden on hospital appointments, thereby contributing to shorter waiting times. Moreover, My IBD Care allows patients to submit PROMs to their clinical teams remotely and in real time, allowing clinical staff to monitor their status and intervene as required.

Scientifically validated digital therapeutics exist for diabetes, cardiovascular disease and sleeping disorders, however there are none addressing the complex, costly challenges of inflammatory conditions.

In the context of these conditions - which include Crohn's, ulcerative colitis, inflammatory arthritis and psoriasis (UK TAM c3.5m people) - a digital therapeutic is digitally-supported behaviour change, tailored to the alleviation of symptoms such as pain, fatigue and anxiety. Importantly, for a therapeutic to be accepted as such, an evidence-based approach is required.

ELIGIBILITY:
Inclusion Criteria:

* • Any patient 16-80 years of age at inclusion

  * Established diagnosis of IBD (including UC, CD, inflammatory bowel disease of uncertain aetiology (IBD-U) and inflammation of an ileo-anal pouch (pouchitis))
  * for more than 6 months prior to enrolment
  * Has a smart phone device with access to the Apple AppStore or Google Play Store
  * On stable medication by which we mean

    * No change in oral 5-ASA dose in the last 1 month. Note, addition of 'as required' topical 5-ASA therapy is permitted
    * Any revent oral corticosteroids must have been finished within 4 weeks. Note
    * No change in immunomodulator dose for 3 months
    * No change in biologic (Adalimumab, Infliximab, Ustekinumab and Vedolizumab) regime for 8 weeks
  * Must be able to comply with all study requirements for the duration of the study as outlined in the protocol.
  * Must be able to understand and be willing to provide written informed consent

Exclusion Criteria:

* • Currently taking part in a clinical trial of an Investigation Medical Procedure

  * Significant psychiatric morbidity
  * Patients likely to change IBD team within the next 12 months
  * Patients taking Cyclosporine or Tacrolimus

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Stable patients with Inflammatory Bowel disease as stipulated above recruited in out-patients and infusion clinics
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year
  Proportion of patients whose care can be maintained via the digital tool through the 12 month period without registering an adverse event:

SECONDARY OUTCOMES:
Health economic assessment | 1 year
  A comparison of the direct and indirect healthcare costs in the 12 month period prior to enrolling in the trial and the 12 month period of the trial
Patient Activation Measure | 1 year
  A comparison of the validated PAM scores at the start and end of the study period
IBD Related Knowledge (CCKNOW) | 1 year
  A comparison of the validated Crohn's and Colitis Knowledge Score at the beginning and end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bu Hayee, PhD, FRCP, Principal Investigator — King's College Hospital NHS Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Selinger CP, Parkes GC, Bassi A, Fogden E, Hayee B, Limdi JK, Ludlow H, McLaughlin S, Patel P, Smith M, Raine T. A multi-centre audit of excess steroid use in 1176 patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2017 Nov;46(10):964-973. doi: 10.1111/apt.14334. Epub 2017 Sep 26. PMID 28949018